CLINICAL TRIAL: NCT03184636
Title: ACLF in Zagazig University Hospitals
Brief Title: Acute-On-Chronic Liver Failure in Zagazig University Hospitals
Acronym: ACLF
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, salem youssef mohamed, assistant professor of internal medicine, gastroenterology and hepatology unit, Zagazig University
Other Study IDs: acute on chronic liver failure
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: ACLF; SOFA; Zagazig university
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale:

To identify the prevalence of Acute-on-chronic liver failure in Zagazig University Hospitals.

The question of the research:

How much the prevalence of Acute-on-chronic Liver Failure in Zagazig University Hospitals?

The aim of the work:

The aim of the study is to identify the presence of Acute-on-chronic Liver Failure in Zagazig University Hospitals

Objectives:

To estimate the prevalence of Acute-on-chronic Liver Failure in Zagazig University Hospitals.

Subjects and Methods:

I . Technical Design:

* Site of the study: Gastroenterology and Hepatology Unit- Zagazig University Hospitals
* Sample size: ''all patients admitted to Gastroenterology and Hepatology Unit with the criteria of ACLF according to EASL-AASLD from June 2017 to December 2017 were included in this study''.

II . OPERATIONAL DESIGN:

* Type of the study: a prospective study.
* Full medical history - taking.
* Full clinical examination.
* Laboratory investigations including Routine laboratory investigation " CBC, Liver functions test, kidney functions test and prothrombin time "

III. Administrative Design:

* Approvals obtained for performing the study from the official or governmental department.
* An ethical committee from the faculty of medicine and patients included in the study.

Results:

Collected data will be presented in tables and suitable graphs and analyzed according to standard statistical methods

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to Gastroenterology and Hepatology Unit with the criteria of ACLF according to EASL-AASLD will be included in this study.

Exclusion Criteria:

* no any exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to Gastroenterology and Hepatology Unit with the criteria of ACLF according to EASL-AASLD will be included in this study.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
improvement of the patients score according to SOFA score (AASLD and EASL guidelines) | 24 weeks from first recruiting
  follow up of participants until the patients recover

SECONDARY OUTCOMES:
death of the patient | 24 weeks from first recruiting
  due to the severity of acute on chronic failure, the death of patients is expected

CONTACTS AND LOCATIONS:
Locations (1):
- Salem Mohamed, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No